CLINICAL TRIAL: NCT07273019
Title: Tongue Muscular Assessment in Children Referred for Polysomnography in a Context of Suspected Obstructive Sleep Apnea
Brief Title: Tongue Muscular Assessment in Children With Sleep Disordered Breathing
Acronym: TMAC-C
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL25_0288; 2025-A01527-42 (Other: ID-RCB)
Record Dates: First submitted 2025-11-19; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: Tongue; Motor functions; Sleep; Sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Polysomnography; Anthropometry; Restraint, Physical

STUDY DESIGN:
Intervention Model Description: Children (4-17 years old) referred to the sleep clinic for polysomnography in a context of suspected obstructive sleep apnea.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children referred for polysomnography for suspected OSA (Experimental): Children aged 4 to 17 years old, referred to the sleep clinic for polysomnography in a context of suspected OSA
  Interventions: Other: Tongue Strength Assessment; Diagnostic Test: Polysomnography; Other: Subjective Assessment of Sleep-Disordered Breathing; Other: Subjective Assessment of Daytime Functioning; Other: Anthropometry; Other: Clinical Examination; Other: Orofacial Praxis Assessment

INTERVENTIONS:
Other: Tongue Strength Assessment — The following items will be assessed:
  1. Tongue peak pressure during 3 seconds of tongue protrusion
  2. Tongue peak pressure (i.e., the maximal pressure - Pmax - exerted against the IOPI bulb) during 3 seconds of tongue elevation
  3. Tongue pressure (in kPa) exerted against the IOPI (Iowa Oral Performance Instrument) bulb while swallowing
Diagnostic Test: Polysomnography — Patients will undergo full-night polysomnography (including the JAWAC system to record mandibular movements) in the sleep unit of Hôpital Femme-Mère-Enfant (Bron, France) to explore OSA.
Other: Subjective Assessment of Sleep-Disordered Breathing — The following questionnaires will be filled out:
  * OSA-18
  * Pediatric Sleep Questionnaire (PSQ)
  * Spruyt & Gozal
  * Sleep Disturbance Scale for Children
  * Abreu et al.'s questionnaire
Other: Subjective Assessment of Daytime Functioning — The following questionnaires will be filled out:
  * Epworth Sleepiness Scale
  * Conners
Other: Anthropometry — The following measures will be collected via the Quick Tongue-Tie Assessment tool:
  1. Maximal mouth opening
  2. Maximal mouth opening with tongue to palate
Other: Clinical Examination — The following variables will be collected during a clinical examination:
  1. Age
  2. Sex
  3. Weight
  4. Height
  5. BMI
  6. Friedman score
  7. Mallampati score
  8. Medical history
Other: Orofacial Praxis Assessment — Bucco-Linguo-Facial Motor Skills will be assessed through the test "Motricité Bucco-Linguo-Faciale" (MBLF).

SUMMARY:
Obstructive sleep apnea (OSA) is part of the sleep-disordered breathing spectrum. Its prevalence in children is 1-5%, and it can have negative consequences at the cardiovascular, cognitive as well as behavioral levels. In children, the first-line treatment is adenotonsillectomy. However, residual obstructive events can persist as the success rate of surgery reaches only 49% in non-obese children. Residual OSA may be explained by multiple sites of obstruction, found in 20-85% children concerned by persistent OSA. Indeed, the tongue appears among one possible primary sites of obstruction. Given the tongue's crucial role in upper-airway patency during sleep, its assessment can inform us about the myofunctional deficits involved in sleep-disordered breathing.

The primary objective of the present study is to assess tongue motor functions in children with sleep-disordered breathing and to compare them to those of healthy children (data collected in a current study (TMAC) conducted at UCLouvain, Belgium; NCT06166680), in order to document possible myofunctional deficits in children with OSA. The hypothesis is that tongue motor functions will be lower in children with sleep-disordered breathing.

ELIGIBILITY:
Inclusion Criteria:

* With suspected sleep-disordered breathing
* Referred for polysomnography
* Affiliated to a social security scheme
* With informed consent from both legal representatives

Exclusion Criteria:

* Insufficient comprehension of French language
* Regarding patients with suspected OSA type I or II:

  * Neurological, cardiac, or respiratory conditions other than sleep disorders and their repercussions
  * Any deficit possibly impacting measurements according to the investigator (e.g., psychiatric condition)
  * Previous surgery performed on the upper airway or the oral cavity
  * Malformation of the skull, the upper airway or the oral cavity
* Regarding patients with suspected OSA type III:

  * Any deficit possibly impacting measurements according to the investigator (e.g., psychiatric condition)
  * Intellectual deficit impeding the understanding of instructions

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-05-17 (Estimated); Study Completion 2027-05-17 (Estimated)

PRIMARY OUTCOMES:
Tongue peak pressure during protrusion | Day 1
  Tongue peak pressure during protrusion will be measured using the IOPI (Iowa Oral Performance Instrument) device. Higher tongue pressure is considered a better outcome.

SECONDARY OUTCOMES:
Tongue peak pressure during elevation and swallowing | Day 1
  Tongue peak pressure during elevation and swallowing movements will be measured using the IOPI (Iowa Oral Performance Instrument) device. Higher tongue pressure is considered a better outcome.
Tongue mobility restriction | Day 1
  Assessed through the ratio between maximal mouth opening and maximal mouth opening with tongue to palate, measured using the Quick Tongue-Tie Assessment tool. Higher values are considered a better outcome.
Orofacial praxis | Day 1
  Orofacial praxis will be assessed through the Motricité Bucco-Linguo-Faciale (MBLF) test, which ranges from 0 to 111. Higher scores indicate a better outcome.
Obstructive apnea-hypopnea index (OAHI) | Day 1
  Respiratory parameters will be assessed by night polysomnography. A higher index indicates a worse outcome.
Central apnea-hypopnea index | Day 1
  Respiratory parameters will be assessed by night polysomnography. A higher index indicates a worse outcome.
Mixed apnea-hypopnea index | Day 1
  Respiratory parameters will be assessed by night polysomnography. A higher index indicates a worse outcome.
Respiratory effort index | Day 1
  Respiratory parameters will be assessed by night polysomnography. A higher index indicates a worse outcome.
Respiratory effort-related arousal index (RERA) | Day 1
  Respiratory parameters will be assessed by night polysomnography. A higher index indicates a worse outcome.
Mean CO2 | Day 1
  Respiratory parameters will be assessed by night polysomnography.
Max CO2 | Day 1
  Respiratory parameters will be assessed by night polysomnography.
Time spent with CO2 > 50mmHg | Day 1
  Respiratory parameters will be assessed by night polysomnography.
Mean SpO2 | Day 1
  Respiratory parameters will be assessed by night polysomnography.
Desaturation index ≥ 3% | Day 1
  Respiratory parameters will be assessed by night polysomnography.
Desaturation index ≥ 4% | Day 1
  Respiratory parameters will be assessed by night polysomnography.
Time spent with SaO2 < 90% | Day 1
  Respiratory parameters will be assessed by night polysomnography.
Total sleep time | Day 1
  Sleep architecture parameters will be assessed by night polysomnography.
Sleep onset latency | Day 1
  Sleep architecture parameters will be assessed by night polysomnography.
Wake after sleep onset | Day 1
  Sleep architecture parameters will be assessed by night polysomnography.
Duration of sleep N1 | Day 1
  Sleep architecture parameters will be assessed by night polysomnography.
Duration of sleep N2 | Day 1
  Sleep architecture parameters will be assessed by night polysomnography.
Duration of sleep N3 | Day 1
  Sleep architecture parameters will be assessed by night polysomnography.
Duration of REM sleep | Day 1
  Sleep architecture parameters will be assessed by night polysomnography.
Sleep efficiency | Day 1
  Sleep architecture parameters will be assessed by night polysomnography.
Score on Abreu's Questionnaire | Day 1
  Total score ranges from 0 to 16. Higher scores indicate a worse outcome.
Score on the OSA-18 Questionnaire | Day 1
  This questionnaire assesses quality of life associated with sleep-disordered breathing in children. Total score ranges from 18 to 126. Higher scores indicate a worse outcome.
Score on the Pediatric Sleep Questionnaire | Day 1
  This questionnaire assesses symptoms and repercussions of sleep-disordered breathing in children. Total score ranges from 0 to 22. Higher scores indicate a worse outcome.
Score on the Spruyt & Gozal Questionnaire | Day 1
  This questionnaire assesses sleep-disordered breathing in children. Total score ranges from 0 to 4. Higher scores indicate a worse outcome.
Score on the Sleep Disturbance Scale for Children | Day 1
  This questionnaire assesses sleep disturbance in children. Total score ranges from 25 to 125. Higher scores indicate a worse outcome.
Score on the French Version of the Sleepiness Scale for Adolescents | Day 1
  This questionnaire assesses excessive daytime sleepiness. Total score ranges from 25 to 125. Higher scores indicate a worse outcome.
Score on the Conners Rating Scale | Day 1
  This questionnaire assesses hyperactivity. Total score ranges from 0 to 30. Higher scores indicate a worse outcome.
Medical history | Day 1
  Medical history is conducted by a doctor. It will be used to determine the type of OSA (craniofacial and/or syndromic comorbidities classify OSA as type III; otherwise, OSA is type II in the presence of obesity, or type I in the absence of obesity).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme-Mère-Enfant : Service d'épileptologie clinique, des troubles du sommeil et de neurologie fonctionnelle de l'enfant, Bron, France

IPD SHARING:
Plan to Share IPD: No